CLINICAL TRIAL: NCT00205166
Title: Does Caffeine Affect the Sensitivity of Adenosine Perfusion Scans?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1999-109
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Coronary Artery Disease
Keywords: adenosine tracer scans; coronary artery disease; caffeine
MeSH Terms: conditions — Coronary Artery Disease | interventions — Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Caffeine 400 mg PO 1 hour before adenosine infusion
  Interventions: Procedure: Cardiac SPECT imaging Rest and Stress; Drug: Caffeine
- 2 (Active Comparator): Caffeine 200 mg po one hour before adenosine infusion
  Interventions: Procedure: Cardiac SPECT imaging Rest and Stress; Drug: Caffeine

INTERVENTIONS:
Procedure: Cardiac SPECT imaging Rest and Stress — adenosine perfusion scintigraphy
Drug: Caffeine — Caffeine 400 mg po
  Arms: 1
Drug: Caffeine — Caffeine 200 mg po
  Arms: 2

SUMMARY:
We are studying the affect of caffeine on the sensitivity of detecting coronary artery disease (blockages in the blood flow to the heart) with adenosine tracer scans. Adenosine is a drug used routinely in patients to relax heart blood vessels in order to assess for the presence of coronary artery disease. Often, if patients have had caffeine, the adenosine scan is not used because of the belief that caffeine may reduce the ability to detect coronary artery disease. We would like to test whether caffeine affects our ability to detect coronary artery disease with adenosine tracer scanning. We will perform an imaging study of the heart with adenosine after you have received caffeine.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have already completed rest/stress 99mTc sestamibi or 99mTc tetrofosmin imaging will be given a form describing this protocol and asked to volunteer for the additional scan

Exclusion Criteria:

* history of asthma, bronchospastic COPD, or renal failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 1999-06; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
This protocol has a specific aim of determining whether prior caffeine administration affects the sensitivity and specificity of adenosine perfusion scintigraphy for detection of impaired coronary vascular reserve. | Assessment is made at the time of research adenosine perfusion scintigraphy

SECONDARY OUTCOMES:
determination of caffeine levels in patients instructed to hold caffeine prior to adenosine imaging | Assess at time of lab sample results obtained

CONTACTS AND LOCATIONS:
Overall Officials: Charles K Stone, MD, Principal Investigator — Univeristy of Wisconsin
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States